CLINICAL TRIAL: NCT00758654
Title: Strain-Encoded Cardiac Magnetic Resonance Imaging as an Adjunct for Dobutamine Stress Testing.
Brief Title: Strain-Encoded Cardiac Magnetic Resonance Imaging for Dobutamine Stress Testing
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, G. Korosoglou, Prof. Dr., Heidelberg University
Other Study IDs: MRI-021
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
Keywords: myocardial strain; Strain-Encoded MRI; dobutamine stress MRI; ischemia; strain rate reserve
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with suspected or known stable coronary artery disease
- 2: Healthy subjects as a control group

SUMMARY:
The purpose of this study is to compare the diagnostic value of SENC to that provided by conventional wall motion analysis for the detection of inducible ischemia during DS-MRI.High-dose dobutamine stress magnetic resonance imaging (DS-MRI) is safe and feasible for the diagnosis of coronary artery disease (CAD) in humans. However, the assessment of cine scans relies on the visual interpretation of regional wall motion, which is subjective. Recently, Strain-Encoded MRI (SENC) has been proposed for the direct color-coded visualization of myocardial strain.

DETAILED DESCRIPTION:
The assessment of inducible regional wall motion abnormalities during high-dose dobutamine stress magnetic resonance imaging (DS-MRI) is an established clinical method with high diagnostic and prognostic value for the evaluation of patients with coronary artery disease (CAD). However, the assessment of cine images relies on the visual interpretation of regional wall motion, which is subjective, and objective approaches for the detection of inducible ischemia with DS-MRI are still lacking.

In our study Strain-Encoded-MRI (SENC) is used for the objective color-coded evaluation of regional myocardial strain during DS-MRI in patients with intermediate to high pretest probability for CAD. We anticipated that this technique would exhibit enhanced sensitivity for the detection of anatomically significant CAD compared to conventional wall motion reading, with invasive coronary angiography used as the standard reference.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or known coronary artery disease

Exclusion Criteria:

* General contraindication for a dobutamine stress or for an MRI examination
* Age < 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with suspected or known coronary artery disease and healthy volunteers serving as a contol group.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Detection of coronary artery disease (>50% diameter stenosis) by invasive angiography | 3 weeks

SECONDARY OUTCOMES:
Long-term mortality and MACE | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Department of Cardiology, Heidelberg, Germany

REFERENCES:
- [Derived] Korosoglou G, Gitsioudis G, Voss A, Lehrke S, Riedle N, Buss SJ, Zugck C, Giannitsis E, Osman NF, Katus HA. Strain-encoded cardiac magnetic resonance during high-dose dobutamine stress testing for the estimation of cardiac outcomes: comparison to clinical parameters and conventional wall motion readings. J Am Coll Cardiol. 2011 Sep 6;58(11):1140-9. doi: 10.1016/j.jacc.2011.03.063. PMID 21884952
- [Derived] Korosoglou G, Lehrke S, Wochele A, Hoerig B, Lossnitzer D, Steen H, Giannitsis E, Osman NF, Katus HA. Strain-encoded CMR for the detection of inducible ischemia during intermediate stress. JACC Cardiovasc Imaging. 2010 Apr;3(4):361-71. doi: 10.1016/j.jcmg.2009.11.015. PMID 20394897